CLINICAL TRIAL: NCT00929422
Title: PET in Evaluating Cerebral Glucose Metabolism and Functional Change for Patients With Spinal Cord Injury
Brief Title: Positron Emission Tomography (PET) in Evaluating Cerebral Glucose Metabolism and Functional Change for Patients With Spinal Cord Injury
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Wang YH, National Taiwan University Hospital
Other Study IDs: 200612018R; NSC 96-2314-B-002-085-MY3
Record Dates: First submitted 2009-06-26; First posted 2009-06-29 (Estimated); Last update posted 2010-12-01 (Estimated); Status verified 2010-11

CONDITIONS: Spinal Cord Injury
Keywords: spinal cord injury; PET; cerebral function; cortical reorganization
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- spinal cord injury 1
- spinal cord injury 2
- spinal cord injury 3
- normal control

SUMMARY:
Background: Spinal cord injury (SCI) results in dysfunction of motor and sensory system and the hormonal secretion. Not only the change of peripheral hormonal organs, the central neurotransmitters were also affected. We consider there are some changes in cerebral physiology, anatomy or function after SCI.

Objective: Use PET imaging to investigate the brain functional difference among the SCI and control group.

DETAILED DESCRIPTION:
Spinal cord injury (SCI) results in dysfunction of motor and sensory system and the hormonal secretion. Not only the change of peripheral hormonal organs, the central neurotransmitters were also affected. We consider there are some changes in cerebral physiology, anatomy or function after SCI. Transcranial magnetic stimulation, magnetic coil or EEG were used to study the phenomenon of cortical reorganization in post-injury of spinal cord. Now functional imaging render the researcher easier to understand adaptive changes of cerebral cortex in patients with SCI. Due to the development of positron emission tomography (PET) and adequate supply of 18-F-deoxyglucose (FDG), the cerebral glucose metabolism and blood flow were approached in easier way. PET was used in patients with cervical compressive myelopathy to evaluate the glucose metabolic rate. Standardized uptake value of FDG and its association with neurological status of pre- and post-operation had been studied. PET was also used to assess the effect of a transverse cord lesion on cerebral energy metabolism in view of sensorimotor reorganization. In addition to FDG, 15O-H2O was applied to evaluate the activation adaptation of post-SCI cerebrum. 13N-NH3 was also used to study the cerebral blood flow by its concentration in brain tissue. Recently the alteration of regional cerebral blood flow was visualized by brain SPECT. We want to know the impact of spinal lesion and function impairment on brain activation in patients with SCI. 6-[18F]fluorodopa (18F-FDOPA) is indicator of brain presynaptic dopaminergic function, which can be used to evaluate the changes of brain dopamine. WE will use 18F-FDOPA-PET to investigate its difference among the SCI and control group.

In our three-year study, 40 men with SCI will be recruited each year, 40 age-matched men as control. In the first year study, FDG-PET will be used to assess the cerebral metabolism, then the glucose metabolic rate of cerebrum and spinal cord will be analyzed. The mechanism of cerebral adaptation after SCI may be clarified. 13N-NH3 will be used in the second year to evaluate the cerebral blood flow in the period of attempted and true action, then their difference will be analyzed by statistical parametric mapping. The picture of activated brain area will be compared between study and control group to investigate the reorganization of cerebral cortex after SCI. In the third year, we will use 18F-FDOPA to evaluate the brain presynaptic dopaminergic function among SCI and control group. Thus, we will delineate the effect of SCI on cerebral function by PET.

ELIGIBILITY:
Inclusion Criteria:

1. age above 18 years old
2. spinal cord injury for over 1 year

Exclusion Criteria:

1. epilepsy
2. psychiatric disorder
3. history of central neurologic system infection
4. Parkinson's disease
5. Alcoholic disease
6. vitamine deficiency

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: right handed patients with spinal cord injury
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2007-08; Primary Completion 2011-08 (Estimated); Study Completion 2011-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Yen-Ho Wang, M.D, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan